CLINICAL TRIAL: NCT04386733
Title: Cardiac Surgery Cancellation at a Large UK Centre and Patient Satisfaction Survey - Quality Improvement Study
Brief Title: Same-day Cardiac Surgery Cancellation
Status: Completed | Type: Observational
Sponsor: St. Bartholomew's Hospital (Other)
Responsible Party: Principal Investigator, Sara Jasionowska, Principal Investigator, St. Bartholomew's Hospital
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Surgery
Keywords: surgery cancellation; cardiac surgery; service improvement; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancelled: all adult patients whose surgery was cancelled on the day of the planned procedure
  Interventions: Other: no intervention, it was an observational study which looked at the reasons for surgical cancellations
- Non-cancelled: all adult patients whose surgery was not cancelled on the day of the planned procedure
  Interventions: Other: no intervention, it was an observational study which looked at the reasons for surgical cancellations

INTERVENTIONS:
Other: no intervention, it was an observational study which looked at the reasons for surgical cancellations — the investigators observed how many patients had their surgeries cancelled and analysed the reasons of these cancellations

SUMMARY:
The investigators prospectively reviewed all same-day cancellations of elective and urgent in-patient adult cardiac surgical procedures from August 2017 to March 2018. Patients were divided into two groups: cancelled (C) and not cancelled (NC). Qualitative patient satisfaction survey was also undertaken.

DETAILED DESCRIPTION:
This prospective audit was performed over a 7-month period (August - March 2018). A quality improvement team, consisting of two clinical research fellows and a consultant cardiothoracic surgeon, reviewed all the cancellations. The research is reported in line with the Standards for Quality Improvement Reporting Excellence (SQUIRE) guidelines.

Adult patients undergoing elective and urgent cardiac surgery were included in our study. Those who underwent emergency or non-cardiac procedures and patients under the age of 18 were excluded. Patients were identified on a weekly basis from theatre registers and printed operating lists. Same day surgery cancellations were defined as any postponement of patients' operation once listed for surgery.

Electronic hospital records were reviewed, and the following information was recorded for all patients: demographics; scheduled surgery date; euroSCORE II and its components; admission type (elective/urgent in-house/transfer patient); date of pre-operative anaesthetic review. Additionally, reasons for cancellation, timing of cancellation (pre-operative/during anaesthesia/intraoperative) and outcomes were recorded. Outcomes included: time from cancellation to performed operation; hospital stay post-cancellation and mortality. Patients were divided into cancelled (C) and non-cancelled (NC) groups for analysis.

The reasons for cancellation were categorized into: lack of ITU beds and nurses; patient medically unfit; scheduling error; patient-related issues; emergency intervened; procedure no longer needed; lack of perfusionist; incomplete investigations; surgeon unavailable; transfer issue; theatre staff shortage; electrical system failure; new intra-operative TOE findings. Patient-related issues included failure to stop medication and treatment refusal. Scheduling errors included overrunning cases, overbooking of the operating room, late operation start and IT errors.

The investigators further assessed the impact of cancellations on patient satisfaction and wellbeing. Patients completed a questionnaire by telephone at 3 months after discharge to allow time to reflect. Questionnaire data assessed adherence to Association of Anaesthetists of Great Britain and Ireland Theatre Efficiency guidance, including healthcare professional informing patients; time offered for explanation; patient understanding and satisfaction as well as perception of being kept nil by mouth (NBM) longer than necessary. (Figure 1) This questionnaire has previously been used by Wasim et al. to assess patient experience following cancelled orthopaedic surgery. A pilot study was conducted to trial the its' validity.

All data was entered into a Microsoft Excel spreadsheet. Statistical analysis consisted of determination of the mean and range for continuous data and percentage quantification for the categorical data. Statistical significance was established using chi-squared test and two-sided unpaired student t-test with p values <0.05 considered significant. The study was approved by the St Bartholomew's Trust Ethics and Quality Improvement Committee. As this was a quality improvement project and information collected did not include personal identifiers, individual consents were not required.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who were scheduled for elective or urgent cardiac surgery

Exclusion Criteria:

* patients under the age of 18 or scheduled for an emergency cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients whose cardiac surgeries were scheduled at the St.Bartholomew's hospital during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1388 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Frequency of cancelled cardiac surgery assessed by number of cancellations | immediately after the cancellation of the same-day surgery
  frequency and reason for same-day cancellations
Reasons for cancellation of cardiac surgery | immediately after the cancellation of the same-day surgery
  reasons for cancelled cardiac surgeries were checked in patients notes and recorded

SECONDARY OUTCOMES:
Patient's satisfaction and reaction to the cancellation assessed by the Patient Satisfaction Questionnaire | throughout study completion, an average of 3 months
  evaluation of patient's reactions to cancellations

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No